CLINICAL TRIAL: NCT00811187
Title: Paracervical Block During Office Hysteroscopy: A Randomized Double Blind Placebo-controlled Trial
Brief Title: Paracervical Block During Office Hysteroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-09-395
Record Dates: First submitted 2008-12-16; First posted 2008-12-18 (Estimated); Results first posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Paracervical Block
Keywords: Hysteroscopy; Pain medication; Lidocaine; Office Procedures
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Lidocaine paracervical block (Experimental): 5cc 1% lidocaine injection in each paracervical region
  Interventions: Drug: Lidocaine paracervical block
- Saline placebo injection (Placebo Comparator): 5cc Normal Saline injection in each paracervical region
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Lidocaine paracervical block — 5cc 1% lidocaine injection in each paracervical region
  Arms: Lidocaine paracervical block
Drug: Normal Saline — 5cc Normal Saline injection in each paracervical region
  Arms: Saline placebo injection

SUMMARY:
The purpose of this study is to determine the effectiveness of paracervical block for pain relief in office hysteroscopy - particularly with the placement of the Essure device. Subjects will be randomized to receive either paracervical block or saline, and will have pain assessments performed throughout the procedure. Subjects and physicians will be blinded to group assignments.

ELIGIBILITY:
Inclusion Criteria:

* Women eligible and scheduled for office hysteroscopic placement of essure devices

Exclusion Criteria:

* Planned secondary procedures
* Lidocaine allergy
* Repeat procedures

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Chudnoff, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Centennial Women's Center / Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Chudnoff S, Einstein M, Levie M. Paracervical block efficacy in office hysteroscopic sterilization: a randomized controlled trial. Obstet Gynecol. 2010 Jan;115(1):26-34. doi: 10.1097/AOG.0b013e3181c51ace. PMID 20027030

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a investigator-sponsored single site clinical trial. Patients were recruited based on physician referral at Montefiore Medical Center from March 2007 to June 2008. Patients were excluded from participation if they had a known allergy to lidocaine.
Pre-assignment Details: Of the 80 patients that met inclusion and exclusion criteria, only 74 completed either the lidocaine or saline placebo single-injection. Patients were randomized 1:1.
Groups:
- Lidocaine Paracervical Block: 10 cc of 1% Lidocaine (10mg) injected in the paracervical region of patient as a single-injection nerve block before their procedure.
- Saline Placebo Injection: 10 cc of Normal Saline (10mg) as placebo injected in paracervical region of patient as a single-injection placebo before their procedure.
Period: Overall Study
Arm/Group | Lidocaine Paracervical Block | Saline Placebo Injection
Started | 40 | 40
Completed | 37 | 37
Not Completed | 3 | 3
Not completed — Unable to place device / procedure abort | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Lidocaine Paracervical Block: 10 cc of 1% Lidocaine injected in the paracervical region
- Saline Placebo Injection: 10 cc of Normal Saline as placebo injected in paracervical region
- Total: Total of all reporting groups
Arm/Group | Lidocaine Paracervical Block | Saline Placebo Injection | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.2 (4.5) | 36.4 (4.1) | 35 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Pain on a 10-point Visual Analog Pain Scale During the Procedure.
Description: This used a visual analog scale from 0 (minimum) to 10 (maximum) that was measured as centimeters. A higher score would indicate more pain, therefore, a worse outcome. Pain was assessed at each step that could potentially elicit pain, specifically when there was direct physical manipulation.
Time Frame: During Procedure
Population: Intent to Treat Population (all participants assigned to lidocaine or saline).
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Lidocaine Group: 10 cc 1% lidocaine injected in the paracervical region
- Saline Placebo Group: 10 cc of 1% lidocaine injected in the paracervical region
Arm/Group | Lidocaine Group | Saline Placebo Group
Number analyzed (Participants) | 37 | 37
Score on a scale | 4.15 (1.9) | 3.38 (5.84)
Statistical Analysis 1: Comparison: Lidocaine Group vs Saline Placebo Group; A sample size calculation and power analysis was conducted using PS Power and Sample Size Calculations 2.1.30 (Vanderbilt University, Department of Biostatistics, Nashville, TN) to determine necessary sample size; Test type: Superiority — [Not Specified]; p < .001, Regression, Linear; Mean Difference (Net) = -2.03 — Treatment pain difference= Lidocaine (0.97) - Placebo (3.00)

ADVERSE EVENTS:
Groups:
- Lidocaine Paracervical Block: 10 cc of 1% (10mg) Lidocaine injected in the paracervical region
- Saline Placebo Injection: 10 cc of Normal Saline (10mg) as placebo injected in paracervical region
Arm/Group | Lidocaine Paracervical Block | Saline Placebo Injection
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/37
Other Adverse Events (participants affected / at risk) | 0/37 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No